CLINICAL TRIAL: NCT03109665
Title: Glaucoma Within Northern Ireland Cohort for the Longitudinal Study of Ageing
Acronym: GwNICOLA
Status: Completed | Type: Observational
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Professor Augusto Azuara-Blanco, Professor, Queen's University, Belfast
Other Study IDs: B16/66
Record Dates: First submitted 2017-03-15; First posted 2017-04-12 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Glaucoma within NICOLA: NICOLA study Participants Eligible for GwNICOLA by meeting inclusion criteria
  Interventions: Diagnostic Test: SD-OCT Angiography; Diagnostic Test: SD-OCT

INTERVENTIONS:
Diagnostic Test: SD-OCT Angiography — SD-OCT Angiography
Diagnostic Test: SD-OCT — SD-OCT

SUMMARY:
Glaucoma is the leading cause of irreversible blindness worldwide. It is caused by damage to the optic nerve between the back of the eye and the brain leading to progressive blindness. The cause is poorly understood but ageing, increased intraocular pressure (IOP) and genetics are all likely to play a role. There is no cure for glaucoma but treatments are available which slow progression. Because vision cannot be restored once lost, early detection, monitoring and early treatment are all essential to preserve visual function.

The condition is diagnosed using a combination of the appearance of the optic nerve on clinical examination or photograph and visual field testing (perimetry). Measurement of IOP and measurement of the thickness of the retinal layers at the back of the eye complement diagnostic decisions.

The Northern Ireland Cohort for the Longitudinal Study of Ageing (NICOLA) study does not include perimetry in the series of tests carried out on all participants but does include photography of the optic nerve, measurement of IOP and measurement of retinal thickness. Therefore we propose to invite back participants of the NICOLA study who have abnormal optic discs and high eye pressure to return for perimetry to confirm a diagnosis of glaucoma. Calling back participants for perimetry is essential to make the diagnosis not only for estimating prevalence but also for identifying participant's ill-health.

The primary aim of this study is to quantify the number of participants in the NICOLA study who have glaucoma and report its risk factors. This will allow an estimate of the number of people in the whole of NI with glaucoma. We will also perform a series of novel tests using state-of-the-art technologies to assess if they are better than current tests at diagnosing glaucoma. This may enable better informed decisions about policy decisions in eyecare.

DETAILED DESCRIPTION:
Purpose and design: This study will answer the following research questions:

1. What is the prevalence of glaucoma within the NICOLA cohort and which systemic and socioeconomic factors influence its prevalence?
2. What is the diagnostic accuracy (sensitivity and specificity) of Retinal Nerve Fibre Layer (RNFL) thickness measurements in the diagnosis of glaucoma?
3. What is the diagnostic accuracy (sensitivity and specificity) of macular thickness analysis in the diagnosis of glaucoma?
4. What is the agreement between intraocular pressure measurement by Ocular Response Analyser (ORA) and Goldmann tonometry?
5. What is the correlation between structural (circumpapillary RNFL or macular Ganglion Cell Complex thickness) or functional measurements (retinal oximetry or perimetry) and Optical Coherence Tomography angiography parameters (% vessel density and vessel calibre) in the assessment of glaucoma?

ELIGIBILITY:
Inclusion Criteria:

1. Participants of the NICOLA study who gave permission to be contacted by the NICOLA study team in future and
2. Vertical cup to disc ratio ≥0.7 and/or inter-eye asymmetry ≥0.2 or neuroretinal rim ≤0.1 or intraocular pressure ≥25 mmHg.

Exclusion Criteria:

1. Non English speakers or
2. Participants of the NICOLA study who did not give permission to be contacted by the NICOLA study team in future

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: NICOLA Study - Random sample of 8500 non-institutionalised adults >50 years from Northern Ireland GwNICOLA participants derived from NICOLA Study
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of Glaucoma in Northern Ireland | 1 day [2 hours]
  Prevalence of Glaucoma in Northern Ireland
Diagnostic Accuracy of Spectral Domain OCT | 1 day [2 hours]
  Diagnostic Accuracy of Spectral Domain OCT

CONTACTS AND LOCATIONS:
Overall Officials: Augusto Azuara-Blanco, PhD, MD, Principal Investigator — Queens University Belfast
Locations (1):
- Northern Ireland Clinical Research Facility, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No